CLINICAL TRIAL: NCT01012973
Title: A Randomized, Double-masked, Sham-controlled Phase 3 Study of the Efficacy, Safety and Tolerability of Repeated Intravitreal Administration of VEGF Trap-Eye in Subjects With Macular Edema Secondary to Central Retinal Vein Occlusion (CRVO)
Brief Title: Vascular Endothelial Growth Factor (VEGF) Trap-Eye: Investigation of Efficacy and Safety in Central Retinal Vein Occlusion (CRVO)
Acronym: GALILEO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14130; 2009-010973-19 (EudraCT Number)
Record Dates: First submitted 2009-10-30; First posted 2009-11-13 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Retinal Vein Occlusion
Keywords: Macular Edema; Central Retinal Vein Occlusion; CRVO; VEGF Trap-Eye; best-corrected visual acuity
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) (Experimental): Participants received a 2 mg dose of Intravitreal Aflibercept Injection (IAI) administered every 4 weeks from Day 1 through Week 20, later as often as every 4 weeks depending on the study retreatment criteria from Week 24 through Week 48. Follow-up phase: Participants on IAI, who continued the study, received 2 mg dose of IAI depending on the study retreatment criteria at Week 60 and 68.
  Interventions: Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321); Other: Sham treatment
- Sham treatment (Sham Comparator): Participants received sham treatment administered every 4 weeks from Day 1 through Week 52. Follow-up phase: Participants on sham treatment, who switched to Intravitreal Aflibercept Injection (IAI), received a 2 mg dose of IAI at week 52 and depending on the study retreatment criteria at Week 60 and 68.
  Interventions: Other: Sham treatment

INTERVENTIONS:
Biological: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) — Intravitreal injection. Weeks 0 to 20 of Aflibercept Injection every 4 weeks; Weeks 24 to 52 every 4 weeks PRN (pro re nata, on demand); plus additional on Week 60 and 68.
  Arms: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321)
Other: Sham treatment — Sham treatment. Weeks 0 to 52 sham treatment every 4 weeks; plus additional on Week 60 and 68.

SUMMARY:
To determine the efficacy of vascular endothelial growth factor (VEGF) Trap-Eye injected into the eye on vision function in subjects with macular edema as a consequence of central retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* Center-involved macular edema secondary to central retinal vein occlusion (CRVO) for no longer than 9 months with mean central subfield thickness ≥ 250 μm on optical coherence tomography (OCT)
* Adults ≥ 18 years
* Early treatment diabetic retinopathy study (ETDRS) best corrected visual acuity (BCVA) of 20/40 to 20/320 (73 to 24 letters) in the study eye

Exclusion Criteria:

* Any prior treatment with anti-VEGF agents in the study eye (Pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc.) or previous administration of systemic anti-angiogenic medications
* Prior panretinal laser photocoagulation or macular laser photocoagulation in the study eye
* CRVO disease duration > 9 months from date of diagnosis
* Previous use of intraocular corticosteroids in the study eye or use of periocular corticosteroids in the study eye within the 3 months prior to Day 1
* Iris neovascularization, vitreous hemorrhage, traction retinal detachment, or preretinal fibrosis involving the macula in either the study eye or fellow eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (61):
- Australia (6):
  - Chatswood, New South Wales
  - Parramatta, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
  - Nedlands, Western Australia
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- France (6):
  - Paris, Cedex 12
  - Nantes, Cedex 1
  - Bordeaux
  - Dijon
  - Marseille
  - Paris
- Germany (24):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Chemnitz, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Kiel, Schleswig-Holstein
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
- Hungary (4):
  - Budapest
  - Debrecen
  - Veszprém
  - Zalaegerszeg
- Italy (8):
  - Ancona
  - Bari
  - Catania
  - Florence
  - Milan
  - Padua
  - Roma
  - Torino
- Japan (5):
  - Nagoya, Aichi-ken
  - Urayasu, Chiba
  - Kyoto, Kyoto
  - Suita, Osaka
  - Chiyoda-ku, Tokyo
- Riga, Latvia
- Singapore, Singapore
- South Korea (3):
  - Seongnam-si, Gyeonggido
  - Incheon
  - Seoul

REFERENCES:
- [Result] Holz FG, Roider J, Ogura Y, Korobelnik JF, Simader C, Groetzbach G, Vitti R, Berliner AJ, Hiemeyer F, Beckmann K, Zeitz O, Sandbrink R. VEGF Trap-Eye for macular oedema secondary to central retinal vein occlusion: 6-month results of the phase III GALILEO study. Br J Ophthalmol. 2013 Mar;97(3):278-84. doi: 10.1136/bjophthalmol-2012-301504. Epub 2013 Jan 7. PMID 23298885
- [Result] Korobelnik JF, Holz FG, Roider J, Ogura Y, Simader C, Schmidt-Erfurth U, Lorenz K, Honda M, Vitti R, Berliner AJ, Hiemeyer F, Stemper B, Zeitz O, Sandbrink R; GALILEO Study Group. Intravitreal Aflibercept Injection for Macular Edema Resulting from Central Retinal Vein Occlusion: One-Year Results of the Phase 3 GALILEO Study. Ophthalmology. 2014 Jan;121(1):202-208. doi: 10.1016/j.ophtha.2013.08.012. Epub 2013 Sep 29. PMID 24084497
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Aflibercept Injection First, Then Aflibercept Injection: Participants received a 2 mg dose of Intravitreal Aflibercept Injection (IAI) administered every 4 weeks from Day 1 through Week 20, later as often as every 4 weeks depending on the study retreatment criteria from Week 24 through Week 48. Follow-up phase: Participants on IAI, who continued the study, received 2 mg dose of IAI depending on the study retreatment criteria at Week 60 and 68.
- Sham Treatment First, Then Aflibercept Injection: Participants received sham treatment administered every 4 weeks from Day 1 through Week 52. Follow-up phase: Participants on sham treatment, who switched to Intravitreal Aflibercept Injection (IAI), received a 2 mg dose of IAI at week 52 and depending on the study retreatment criteria at Week 60 and 68.
Period: Overall Study
Arm/Group | Aflibercept Injection First, Then Aflibercept Injection | Sham Treatment First, Then Aflibercept Injection
Started | 106 | 71
Participants Received Treatment | 104 (Safety Population: Participants received treatment) | 68 (Safety Population: Participants received treatment)
Fulfilled Requirements of FAS Population | 103 (Full Analysis Set (FAS) Population: Participants received treatment with post baseline measurements) | 68 (Full Analysis Set (FAS) Population: Participants received treatment with post baseline measurements)
Completed Week 24, From FAS | 97 | 57
Completed Week 52, From FAS | 91 | 52
Completed | 90 | 52
Not Completed | 16 | 19
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 0 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — (Overseas travel - indefinite period) | 1 | 0
Not completed — Increase in vis. acuity, never injected | 0 | 1
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment | Total
Number analyzed (Participants) | 104 | 68 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (12.3) | 63.8 (13.3) | 61.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 31 | 76
  Male | 59 | 37 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 100 | 66 | 166
  Unknown or Not Reported | 0 | 1 | 1
Baseline Best Corrected Visual Acuity (BCVA) letter scores [Mean (Standard Deviation); unit: Letters correctly read] — Infiormation retrieved from all baseline participants. Only participants with a ETDRS (Early Treatment Diabetic Retinopathy Study) Best Corrected Visual Acuity letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye at 4 meters were included; a higher score represents better functioning.
  Letters correctly read | 53.5 (15.7) | 50.9 (15.4) | 52.5 (15.6)
Number of participants with baseline retinal perfusion [Number; unit: Participants] — Retinal perfusion defined as less than 10 disc areas of capillary nonperfusion using fluorescein angiography (FA)
  Participants
    Perfused | 90 | 54 | 144
    Nonperfused | 7 | 7 | 14
    Indeterminate | 7 | 7 | 14
Baseline Retinal Thickness by Optical Coherence Tomography (OCT) [Mean (Standard Deviation); unit: microns] | 682.78 (233.36) | 638.66 (224.69) | 665.34 (230.33)
Baseline intraocular pressure [Mean (Standard Deviation); unit: mm Hg] | 15.2 (2.8) | 14.4 (2.7) | 14.9 (2.8)
Number of participants with time since Central retinal vein occlusion (CRVO) diagnosis [Number; unit: Participants]
  >= 2 months | 46 | 33 | 79
  < 2 months | 56 | 35 | 91
  Missing | 2 | 0 | 2
Baseline National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) total score [Mean (Standard Deviation); unit: scores on a scale] — The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
  scores on a scale | 79.66 (13.06) | 78.94 (14.00) | 79.38 (13.40)
European questionnaire 5 dimensions (EQ-5D) total score [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D total score ranges from -0.594 to 1.000 with -0.594 being the worst.
  score on a scale | 0.87 (0.15) | 0.86 (0.16) | 0.87 (0.15)
Race [Number; unit: Participants]
  Asian | 26 | 15 | 41
  White | 75 | 49 | 124
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 24 With Discontinued Participants Before Week 24 Evaluated as Failures
Description: Defined study baseline range of Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score of 73 to 24 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning. Nominator = (Number of participants who maintained vision * 100); Denominator = Number of participants analyzed.
Time Frame: Baseline and Week 24
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 103 | 68
Percentage of participants | 60.2 | 22.1
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Null hypothesis of difference of Eylea minus Sham of 0 was tested. In the database close after Week 24, basis for primary efficacy evaluation, 56 Sham / 96 Eylea subjects were considered as week 24 completers; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 38.3, 95% CI 2-sided [24.4 to 52.1] — The estimate is calculated as Eylea minus Sham. A positive value shows Eylea showed a higher BCVA total score compared to Sham

2. Secondary Outcome: Change From Baseline in BCVA as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 24 - Last Observation Carried Forward (LOCF)
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity letter score of 73 to 24 (= Acuity of 20/40 to 20/320) in the study eye; a higher score represents better functioning. However, because this was assessed at the screening visit, subjects may have had a higher BCVA recorded at the baseline visit and would not have been excluded from the study.
Time Frame: Baseline and Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 103 | 68
Letters correctly read | 71.6 (17.1) | 54.3 (20.2)
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Null hypothesis was equality in change from baseline to Week 24 in BCVA total letter score between Eylea and Sham. If primary efficacy was successful, secondary efficacy endpoints were tested in a pre-specified fixed sequence testing procedure. Change in BCVA letter score was to be tested first in this sequence; Test type: Superiority or Other; p < .0001, ANOVA — As primary efficacy evaluation was significant, and this p-value was below significance level of two-sided <.05, the fixed sequence testing did continue with next secondary endpoint; ANOVA, adjusting for region and baseline BCVA category as fixed factors; Difference in Least square means = 14.7, 95% CI 2-sided [10.8 to 18.7] — The difference is calculated as Eylea minus Sham. A positive value indicates Eylea showed a higher change in BCVA total score until week 24 compared to Sham

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 24 - LOCF
Time Frame: Baseline and Week 24
Population: Full-Analysis Set with assessment for this outcome measure; imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 103 | 67
microns | -448.58 (256.02) | -169.27 (224.72)
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Null hypothesis was equality in change from baseline to Week 24 in central retinal thickness between Eylea and Sham. If primary efficacy was successful, secondary efficacy end points were to be tested in a pre-specified fixed sequence testing procedure. Change in central retinal thickness was to be tested at second place in this sequence; Test type: Superiority or Other; p < .0001, ANCOVA — As fixed sequence testing did reject nullhypothesis of change from baseline in BCVA until week 24, and this p-value was below significance level of two-sided <.05, the fixed sequence testing did continue with next secondary endpoint; ANCOVA, stratified by region and baseline BCVA category, baseline central retinal thickness added as covariate; Difference in Least square (LS) means = -239.42, 95% CI 2-sided [-286.31 to -192.53] — The difference is calculated as Eylea minus Sham. A negative value indicates Eylea showed a higher reduction in change in central retinal thickness until week 24 compared to Sham

4. Secondary Outcome: Percentage of Participants Who Developed Neovascularization During the First 24 Weeks
Description: Formation of blood vessels in the anterior segment, optic disc, or elsewhere in the fundus up to Week 24
Time Frame: From baseline until Week 24
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 103 | 68
Percentage of participants
  Any neovascularization | 2.9 | 4.4
  Anterior segment neovascularization | 1.9 | 1.5
  Neovascularization of the optic disc (NVD) | 0.0 | 0.0
  Neovascularization elsewhere in the fundus (NVE) | 1.0 | 2.9
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Nullhypothesis of no difference in development of neovascularizations between Eylea and Sham group was tested. (Any neovascularization); Test type: Superiority or Other; p = 0.5947, Cochran-Mantel-Haenszel — As fixed sequence testing did reject nullhypothesis of change from baseline in CRT until week 24, and this p-value was not below significance level of two-sided <.05, the fixed sequence testing did end with this evaluation; Cochrane-Mantel-Haenszel test, stratified by region and baseline BCVA category; CMH adjusted Difference = -1.5, 95% CI 2-sided [-7.4 to 4.4]

5. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score at Week 24 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight
Time Frame: Baseline and Week 24
Population: Full-Analysis Set with assessment for this outcome measure; imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 96 | 65
Scores on a scale | 7.46 (9.55) | 3.55 (9.74)
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Test type: Superiority or Other; Difference in LS means = 4.2, 95% CI 2-sided [1.7 to 6.8] — As the fixed sequence of secondary endpoints stopped with proportion of neovascularizations developed until week 24, 95% confidence interval is only of descriptive nature

6. Secondary Outcome: Change From Baseline in European Five-dimensional Health Scale (EQ-5D) Score at Week 24 - LOCF
Description: EQ-5D is a quality of life questionnaire based on a scale from -0.594 (worst) to 1.00 (best).
Time Frame: Baseline and Week 24
Population: Full-Analysis Set with assessment for this outcome measure; imputation technique: LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | Sham Treatment
Number analyzed (Participants) | 95 | 64
Scores on a scale | 0.029 (0.139) | -0.002 (0.195)
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs Sham Treatment; Test type: Superiority or Other; Difference in LS Means = 0.044, 95% CI 2-sided [-0.002 to 0.09] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Groups:
- Aflibercept Injection (Until Week 20): Participants received a 2 mg dose of Intravitreal Aflibercept Injection (IAI) administered every 4 weeks from Day 1 through Week 20. Participants were observed until Week 24. Participants in the safety population were at risk.
- Sham Treatment (Until Week 20): Participants received sham treatment administered every 4 weeks from Day 1 through Week 20. Participants were observed until Week 24. Participants in the safety population were at risk.
- Aflibercept Injection (Until Week 48): Participants who continued the study drug until Week 24 received a 2 mg dose of Intravitreal Aflibercept Injection (IAI) administered as often as every 4 weeks depending on the study retreatment criteria from Week 24 through Week 48. Participants were observed from Week 24 until Week 52. Participants in the safety population that completed Week 24 were at risk.
- Sham Treatment (Until Week 48): Participants who continued the study drug until Week 24 received sham treatment administered every 4 weeks from Week 24 to Week 48. Participants were observed from Week 24 until Week 52. Participants in the safety population that completed Week 24 were at risk.
- Aflibercept Injection Continued (Until Week 68): Participants on IAI who continued the study drug until Week 52, received 2 mg dose of IAI depending on the study retreatment criteria at Week 52, 60 and 68. Participants were observed starting from Week 52. Participants in the safety population that completed Week 52 were at risk.
- Sham Treatment Then Aflibercept Injection (Until Week 68): Participants on sham treatment switched to IAI, received a 2 mg dose of IAI at Week 52 and depending on the study retreatment criteria at Week 60 and 68. Participants were observed starting from Week 52. Participants in the safety population that completed Week 52 were at risk.
Arm/Group | Aflibercept Injection (Until Week 20) | Sham Treatment (Until Week 20) | Aflibercept Injection (Until Week 48) | Sham Treatment (Until Week 48) | Aflibercept Injection Continued (Until Week 68) | Sham Treatment Then Aflibercept Injection (Until Week 68)
Serious Adverse Events (participants affected / at risk) | 8/104 | 8/68 | 14/97 | 7/57 | 4/91 | 3/52
Other Adverse Events (participants affected / at risk) | 52/104 | 44/68 | 66/97 | 30/57 | 38/91 | 19/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection (Until Week 20) (N=104) | Sham Treatment (Until Week 20) (N=68) | Aflibercept Injection (Until Week 48) (N=97) | Sham Treatment (Until Week 48) (N=57) | Aflibercept Injection Continued (Until Week 68) (N=91) | Sham Treatment Then Aflibercept Injection (Until Week 68) (N=52)
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Iris neovascularisation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Macular ischaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 2 | 4 | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0 | 2 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic heart disease prophylaxis (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection (Until Week 20) (N=104) | Sham Treatment (Until Week 20) (N=68) | Aflibercept Injection (Until Week 48) (N=97) | Sham Treatment (Until Week 48) (N=57) | Aflibercept Injection Continued (Until Week 68) (N=91) | Sham Treatment Then Aflibercept Injection (Until Week 68) (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 10 | 3 | 3 | 0 | 9 | 3
Eye irritation (Eye disorders) | 3 | 7 | 4 | 1 | 1 | 2
Eye pain (Eye disorders) | 12 | 3 | 6 | 2 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 6 | 5 | 2 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 3 | 4 | 3 | 4 | 1 | 2
Macular fibrosis (Eye disorders) | 1 | 1 | 5 | 4 | 0 | 3
Macular ischaemia (Eye disorders) | 7 | 5 | 3 | 1 | 0 | 1
Macular oedema (Eye disorders) | 2 | 9 | 30 | 7 | 17 | 2
Ocular hyperaemia (Eye disorders) | 5 | 4 | 2 | 1 | 4 | 1
Optic disc vascular disorder (Eye disorders) | 5 | 3 | 3 | 3 | 0 | 0
Retinal exudates (Eye disorders) | 8 | 5 | 4 | 3 | 0 | 0
Retinal haemorrhage (Eye disorders) | 4 | 6 | 11 | 5 | 5 | 2
Retinal vascular disorder (Eye disorders) | 6 | 7 | 10 | 2 | 0 | 2
Visual acuity reduced (Eye disorders) | 2 | 7 | 10 | 1 | 7 | 1
Vitreous detachment (Eye disorders) | 2 | 1 | 7 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 6 | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 5 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 8 | 6 | 10 | 11 | 4 | 2
Intraocular pressure increased (Investigations) | 9 | 4 | 14 | 2 | 2 | 1
Visual acuity tests abnormal (Investigations) | 0 | 1 | 5 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 7 | 4 | 4 | 1 | 1 | 1
Hypertension (Vascular disorders) | 4 | 3 | 4 | 4 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publishing of result communication only after Bayer´s written approval. Manuscript to Bayer sixty days before public release. If no written Bayer comment within 60 days consider approval given. If multi-site study, principal investigator (PI) not do independently publish results before publication of the multi-site paper, but PI not restricted from 24 months from study to completion onwards.